CLINICAL TRIAL: NCT06183606
Title: Local Antibiotic Prophylaxis With Antibiotic Cement: Interest of High-dose Gentamicin Cement Associated With Clindamycin in Changes of Hip and Knee Prostheses
Brief Title: Interest of High-dose Gentamicin Cement Associated With Clindamycin in Changes of Hip and Knee Prostheses
Acronym: HKP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7411
Record Dates: First submitted 2022-10-26; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Hip or Knee Replacement
Keywords: Hip Replacement; knee Replacement; Local antibiotic prophylaxis; Antibiotic cement; Gentamicin cement; Clindamycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A hip or knee prosthesis can be cemented or not. The team of orthopedic surgeons from the CCOM (Centre de Chirurgie Orthopédique et de la Main) has been cementing all hip and knee prosthesis poses for many years using gentamycin cement as recommended by the French Society of Orthopedic Surgery. and trauma (SOFCOT) (1). Data obtained from the Norwegian Register of Hip Prostheses show that the best survival curve for these prostheses is found for prostheses cemented with gentamycin cement (all causes combined). Independently of the risk of aseptic loosening, infection on the prosthesis is the second complication of arthroplasty. The defense mechanism against pathogens in contact with an implant is the formation of a biofilm. Biofilm bacteria are metabolically inactive and characterized by stationary growth. Due to their slower replication, bacteria in biofilm are up to 1000 times more resistant to antibiotics. Therefore, the optimization of local antibiotic prophylaxis is essential.

ELIGIBILITY:
Inclusion criteria:

* Adult subject (≥18 years old)
* Patient operated on at the HUS between 01/02/2017 and 31/01/2019, for replacement of hip and knee prostheses
* Patient having given their consent for the reuse of their data for the purposes of this research

Exclusion criteria:

- Patient who expressed their opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥18 years old) operated on at the HUS between 01/02/2017 and 31/01/2019, for replacement of hip and knee prostheses.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-06-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of surgical site infections (SSI) after changes of hip and knee prostheses | Through study completion, an average of 3 months
  Retrospective description of the benefit of high-dose gentamicin cement combined with clindamycin in hip and knee prosthesis changes

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique Septique - CHU de Strasbourg - France, Strasbourg, France